CLINICAL TRIAL: NCT02838706
Title: Contionuous Perioperative Hemoglobin and Perfusion Index Measurements in Elderly Patients With Hip Fracture and Post Operative Delirium
Brief Title: Elderly With Hip Fracture and Perioperative Hemoglobin and Perfusion Index Levels
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christopher Clemmesen, MD, Hvidovre University Hospital
Other Study IDs: HvidovreUH
Record Dates: First submitted 2016-04-18; First posted 2016-07-20 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Anemia; Delirium
Keywords: postoperative anemia; perfusion index
MeSH Terms: conditions — Anemia; Delirium | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elderly with hip fracture: The subjects are patients age ≥ 65 years requiring surgery for a hip fracture
  Interventions: Procedure: Surgery for hip fracture

INTERVENTIONS:
Procedure: Surgery for hip fracture

SUMMARY:
The overall aim of the study is to investigate the time difference in the diagnosing of anemia among elderly with hip fracture, between measurements with standard blood samples and non-invasive SpHb-measuring. Another aim is to investigate the relationship between perfusion index and prolong perioperative anemia and the potential impact on perioperative complications.

DETAILED DESCRIPTION:
Immediately after admission and diagnosis of a hip fracture the patients will be monitored with Masimo SpHb. The Patients will be continuously measured until the third day after surgery. The Monitors Hb and PI data but not the SpO2% will be blinded to all participating healthcare personnel.The first three postopertive days the patiens will daily be examined to determined it they have developed delirium.

All perioperativ complications in that period will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Primary hip fracture requiring surgery
* Patients able to give informed consent
* Patients who are able to undergo the Hospitals standardized fast track
* Perioperative care regimen for hip fracture including are pre operative placed epidural

Exclusion Criteria:

* Patients who can not co-operate to have a sensor attach to the finger continuous for 4 days.
* Patients who has allergy to the bandage that is used to attach the sensor.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The subjects are patients age ≥ 65 years requiring surgery for a hip fracture.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Delay in diagnosting perioperative anemia | From admission up to and including the 3 postopertive day
  Description of lag time between detection of anaemia by SpHb and Hb by blood sampling/transfusion
Perfusion index, periopertive anemia and delirium | From admission up to and including the 3 postopertive day
  The relation between average perioperative perfusion index, cumulated perioperative anemia over time and patient outcome in the form of medical complications, mortality, delirium and LOS.

SECONDARY OUTCOMES:
Perfusion index as a predictor of early warning score (EWS) | From admission up to and including the 3 postopertive day
  Is there a relationship between low perfusion index an high EWS?

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Hvidovre, department of anesthesiology, Hvidovre, Denmark